CLINICAL TRIAL: NCT02187523
Title: Relative Oral Bioavailability of 40 mg Telmisartan / 12.5 mg HCTZ Fixed Dose Combination Compared With Its Monocomponents in Healthy Subjects. A 4 Period Cross-over, Open, Randomized, Replicate Design Study
Brief Title: Relative Oral Bioavailability of Telmisartan / Hydrochlorothiazide (HCTZ) Fixed Dose Combination (FDC) Compared With Its Monocomponents in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.324
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrochlorothiazide; Telmisartan

ARMS (2):
- Telmisartan/HCTZ FDC (Experimental)
  Interventions: Drug: Telmisartan/HCTZ FDC
- Telmisartan and HCTZ individual tablets (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide; Drug: Telmisartan

INTERVENTIONS:
Drug: Hydrochlorothiazide
  Arms: Telmisartan and HCTZ individual tablets
Drug: Telmisartan
  Arms: Telmisartan and HCTZ individual tablets
Drug: Telmisartan/HCTZ FDC
  Arms: Telmisartan/HCTZ FDC

SUMMARY:
A study to demonstrate the bioequivalence of telmisartan and HCTZ administered as fixed dose combination in comparison to the single unit formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 55 years
* Broca ≥ -20 % and ≤ +20 %

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Supine blood pressure at screening of systolic ≤ 110 mmHg and diastolic ≤ 60 mmHg
* History of orthostatic hypotension, fainting, spells or blackouts
* Chronic or relevant acute infection
* History or allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) ≤ 1 month prior to administration or during the trial
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation (≤ 1 month prior to administration or during the trial)
* Excessive physical activities (≤ 5 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Hypersensitivity to Telmisartan and/or HCTZ and/or related classes of drugs

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (e.g. sterilization, intrauterine device (IUD), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 1999-10; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Total area under concentration-time curve of the analytes in plasma from time zero to infinity (AUC0-∞) | Pre-dose up to day 54
Maximum concentration of the analytes in plasma (Cmax) | Pre-dose up to day 54
Amount of HCTZ excreted in urine over 48 h (Ae(0-48)) | Pre-dose up to day 50

SECONDARY OUTCOMES:
time to achieve maximum concentration of the analytes in plasma (tmax) | Pre-dose up to day 54
Terminal elimination half life of the analytes in plasma (t1/2) | Pre-dose up to day 54
Total clearance of the of the analytes after oral administration (CLtot/f) | Pre-dose up to day 54
Total mean residence time of the analytes (MRTtot) | Pre-dose up to day 54
Apparent volume of distribution of the analytes during the terminal phase (Vz/f) | Pre-dose up to day 54
Number of patients with relevant changes in laboratory values | Screening (day -14 to day 0) and day 72
Number of patients with relevant changes in vital signs (blood pressure, pulse rate) | Up to day 72
Number of patients with Adverse events | Up to day 72
Number of patients with relevant changes in ECG | Screening (day -14 to day 0) and day 72
Number of patients with relevant changes in physical examination | Screening (day -14 to day 0) and day 72